CLINICAL TRIAL: NCT06798012
Title: A Phase 2, Open-label, Proof-of-Concept Study to Investigate the Efficacy, Safety, and Tolerability of TAK-411 in Adult Subjects With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (The CASCA Study)
Brief Title: A Study of TAK-411 in Adults With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Acronym: CASCA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-411-2001
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Keywords: Drug Therapy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-411 (Experimental): Participants will receive TAK-411 400 milligrams per kilogram (mg/kg), IV infusion as an induction dose on Day 1 of initial treatment period. The induction dose may be repeated once after 3 weeks if participants exhibit no clinical change. Thereafter, participants will receive TAK-411 200 mg/kg, IV infusion every 3 weeks for a total of 24 weeks (initial treatment period), followed by an optional additional 27 weeks (extended treatment period).
  Interventions: Biological: TAK-411

INTERVENTIONS:
Biological: TAK-411 — TAK-411 IV infusion.
  Other Names: Hypersialylated Immune Globulin G

SUMMARY:
CIDP is an autoimmune disease. This means that the body's germ fighting (immune) system attacks itself. In CIDP, the immune system attacks the protective covering around the nerves called myelin. Over time, these nerves lose their ability to send signals to the muscles in the body. This leads to muscle weakness and loss of sensation in arms and legs among other symptoms. Participants with CIDP can be treated with a protein called immunoglobulin (or IG).

TAK-411 is a special type of immune globulin G (hsIgG) that has been chemically changed. It is made from IG that comes from human plasma. This study will test if TAK-411 can decrease inflammation and improve symptoms of CIDP.

The main aim of this study is to check how TAK-411 affects the physical functioning of adults with CIDP when compared with results of the placebo group of a historical trial.

Participants may be treated with TAK-411 for up to 1 year (51 weeks) and will be followed up for 3 weeks after last dose.

During the study, participants may visit their study clinic up to approximately 21 times.

ELIGIBILITY:
Key Inclusion Criteria

* The participant is at least 18 years of age, inclusive, at the time of signing the Informed Consent Form (ICF).
* The participant has a body weight of less than or equal to (<=) 150 kilogram (kg).
* The participant has a documented diagnosis of typical CIDP, as confirmed by a neurologist specializing/experienced in neuromuscular diseases and consistent with the European Academy of Neurology/Peripheral Nerve Society (EAN/PNS) 2021 criteria.
* The participant has responded to IgG treatment in the past (documented partial or complete resolution of neurological symptoms and deficits).
* The participant has had disease activation within 18 months before screening, as documented in medical records and in the opinion of the investigator, defined as one of the following:

  1. Clinically meaningful deterioration of symptoms on interruption or dose reduction of IgG treatment.
  2. Clinically meaningful deterioration of symptoms requiring IgG treatment dose increase with subsequent clinical improvement.
  3. Clinically meaningful deterioration of symptoms at the end of IgG treatment dose interval with improvement after next dose administration.
* The participant is on a stable dose of immunoglobulin treatment intravenously (IGIV) treatment, defined as no change greater than 10 percentage (%) in frequency or dose of IGIV therapy within the 12 weeks before and throughout screening within the dose range of 0.4 to 2.4 grams per kilogram (g/kg) every 2 to 6 weeks (inclusive).
* The participant has an INCAT score greater than (>) 2 at screening.

Key Exclusion Criteria

* The participant has a documented diagnosis of a CIDP variant per EAN/PNS 2021 criteria.
* The participant has any neuropathy of other causes, including the following:

  1. Hereditary demyelinating neuropathies, such as hereditary sensory and motor neuropathy, Charcot-Marie-Tooth disease, and hereditary sensory and autonomic neuropathies.
  2. Neuropathies secondary to infections, disorders, or systemic diseases such as Borrelia burgdorferi infection (Lyme disease), diphtheria, systemic lupus erythematosus, POEMS (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes) syndrome, osteosclerotic myeloma, diabetic and nondiabetic lumbosacral radiculoplexus neuropathy, lymphoma, amyloidosis.
  3. Multifocal motor neuropathy.
  4. Drug-, biologic-, chemotherapy-, or toxin-induced peripheral neuropathy.
  5. Diabetic peripheral neuropathy.
* The participant has any chronic or debilitating disease, or central nervous disorder that causes neurological symptoms or that may interfere with assessment of CIDP or outcome measures, including (but not limited to) multiple sclerosis, arthritis, stroke, and Parkinson's disease.
* The participant is required to take or has taken immunomodulatory/immunosuppressive agents (except IGIV) that include, but are not limited to, complement inhibitors, rituximab, efgartigimod, and chemotherapeutic drugs, within 6 months of screening.
* The participant has undergone plasma exchange within 3 months of screening.
* The participant has a history of malignancy with less than 2 years of complete remission before screening, or active malignancy requiring chemotherapy and/or radiotherapy.

Note: Participants with adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or stable prostate cancer not requiring treatment are eligible.

* The participant has experienced deep vein thrombosis or arterial thromboembolic events (example, cerebrovascular accident, pulmonary embolism) within 12 months of screening.
* The participant has any medical condition, laboratory finding, or physical examination finding that precludes participation or with clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may interfere with successful completion of the study or place the participant at undue medical risk.
* The participant has participated in another clinical study involving an IP or investigational device within 30 days before screening or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-12-02 (Estimated); Study Completion 2028-06-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Improvement in Functional Ability at Week 24 | At Week 24
  Improvement in functional ability is defined as decrease of >=1 point in INCAT score at Week 24 compared with baseline (last assessment before first investigational product [IP] administration on Day 1). INCAT disability scale consists of upper and lower extremity components, which are scored based on a participant's level of impairment/disability in their arms and legs, respectively. Each component is scored from 0 to 5 points, which are summed for an overall INCAT disability score ranging from 0 to 10 points, where a score of 0 indicates no signs of disability (example, no upper limb problems and walking not affected) and a score of 10 indicates most severe disability (example, inability to move either arm for any purposeful movement and restricted to a wheelchair, unable to stand and walk a few steps with help). Adjusted INCAT disability score remains identical to INCAT disability score, except that changes in upper limb function from 0 (normal) to 1 (minor symptoms) are excluded.

SECONDARY OUTCOMES:
Number of Participants With Improvement in Functional Ability at Weeks 12 and 54 | At 12 and 54 weeks
  Improvement in functional ability is defined as decrease of >=1 point in the adjusted INCAT score at 12 and 54 weeks compared with baseline (last assessment before first IP administration on Day 1). INCAT disability scale consists of upper and lower extremity components, which are scored based on a participant's level of impairment/disability in their arms and legs, respectively. Each component is scored from 0 to 5 points, which are summed for an overall INCAT disability score ranging from 0 to 10 points, where a score of 0 indicates no signs of disability (example, no upper limb problems and walking not affected) and a score of 10 indicates most severe disability (example, inability to move either arm for any purposeful movement and restricted to a wheelchair, unable to stand and walk a few steps with help). Adjusted INCAT disability score remains identical to INCAT disability score, except that changes in upper limb function from 0 (normal) to 1 (minor symptoms) are excluded.
Change From Baseline in Adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) Score | Baseline (last assessment prior first dose on Day 1), at 12, 24 and 54 weeks
  INCAT disability scale consists of upper and lower extremity components, which are scored based on a participant's level of impairment/disability in their arms and legs, respectively. Each component is scored from 0 to 5 points, which are summed for an overall INCAT disability score ranging from 0 to 10 points, where a score of 0 indicates no signs of disability (example, no upper limb problems and walking not affected) and a score of 10 indicates most severe disability (example, inability to move either arm for any purposeful movement and restricted to a wheelchair, unable to stand and walk a few steps with help). Adjusted INCAT disability score remains identical to INCAT disability score, except that changes in upper limb function from 0 (normal) to 1 (minor symptoms) are excluded.
Change From Screening in the Adjusted INCAT Score | Screening, at 12, 24 and 54 weeks
  INCAT disability scale consists of upper and lower extremity components, which are scored based on a participant's level of impairment/disability in their arms and legs, respectively. Each component is scored from 0 to 5 points, which are summed for an overall INCAT disability score ranging from 0 to 10 points, where a score of 0 indicates no signs of disability (example, no upper limb problems and walking not affected) and a score of 10 indicates most severe disability (example, inability to move either arm for any purposeful movement and restricted to a wheelchair, unable to stand and walk a few steps with help). Adjusted INCAT disability score remains identical to INCAT disability score, except that changes in upper limb function from 0 (normal) to 1 (minor symptoms) are excluded.
Number of Participants With Improvement in Functional Ability on Inflammatory Rasch-built Overall Disability Scale (I-RODS) Score | At 12, 24 and 54 weeks
  Improvement in functional ability defined as increase of greater than or equal to (>=) 4 points in the raw summed I-RODS score at 12, 24, and 54 weeks compared with baseline. I-RODS is a validated, participants-reported, linearly weighted overall disability scale that was specifically designed to capture current activity and social participation limitations in participants with immune-mediated peripheral neuropathies including CIDP. I-RODS comprises 24 items for which participants are asked to rate their functioning related to a variety of everyday tasks at the moment of completion. The participant assigns a score between 0 and 2 to each item as follows:0 (impossible to perform),1 (performed with difficulty), 2 (easily performed) with a lower score indicating more severe activity and social participation limitations. A total I-RODS score of 0 (complete disability) to 48 (no disability) is tabulated by totalling the 24-item responses where higher score represents better outcomes.
Change From Baseline in I-RODS Score | Baseline (last assessment prior first dose on Day 1), at 12, 24 and 54 weeks
  The I-RODS is a validated, participants-reported, linearly weighted overall disability scale that was specifically designed to capture current activity and social participation limitations in participants with immune-mediated peripheral neuropathies including CIDP. The I-RODS comprises 24 items for which participants are asked to rate their functioning related to a variety of everyday tasks at the moment of completion. The participant assigns a score between 0 and 2 to each item as follows: 0 (impossible to perform), 1 (performed with difficulty), 2 (easily performed) with a lower score indicating more severe activity and social participation limitations. A total I-RODS score of 0 (complete disability) to 48 (no disability) is tabulated by totalling the 24-item responses where higher score represents better outcomes.
Change From Screening in I-RODS Score | Screening, at 12, 24 and 54 weeks
  The I-RODS is a validated, participants-reported, linearly weighted overall disability scale that was specifically designed to capture current activity and social participation limitations in participants with immune-mediated peripheral neuropathies including CIDP. The I-RODS comprises 24 items for which participants are asked to rate their functioning related to a variety of everyday tasks at the moment of completion. The participant assigns a score between 0 and 2 to each item as follows: 0 (impossible to perform), 1 (performed with difficulty), 2 (easily performed) with a lower score indicating more severe activity and social participation limitations. A total I-RODS score of 0 (complete disability) to 48 (no disability) is tabulated by totalling the 24-item responses where higher score represents better outcomes.
Change From Baseline in Medical Research Council Sum Score (MRC-SS) | Baseline (last assessment prior first dose on Day 1), at 12, 24 and 54 weeks
  The MRC-SS is used clinician-reported measure of muscle strength. Assessments are conducted bilaterally on six muscle groups: upper arm abductors, elbow flexors, wrist extensors, hip flexors, knee extensors, and foot dorsal flexors. Each muscle is rated from 0 to 5, where 0 indicates no visible contraction and 5 indicates normal strength. The scores are summed to obtain the MRC-SS, which ranges from 0 (quadriplegic) to 60 (normal strength).
Change From Screening in MRC-SS | Screening, at 12, 24 and 54 weeks
  The MRC-SS is used clinician-reported measure of muscle strength. Assessments are conducted bilaterally on six muscle groups: upper arm abductors, elbow flexors, wrist extensors, hip flexors, knee extensors, and foot dorsal flexors. Each muscle is rated from 0 to 5, where 0 indicates no visible contraction and 5 indicates normal strength. The scores are summed to obtain the MRC-SS, which ranges from 0 (quadriplegic) to 60 (normal strength).
Change From Baseline in Bilateral Hand Grip Strength | Baseline (last assessment prior first dose on Day 1), at 12, 24 and 54 weeks
  Bilateral hand grip strength assessments will be performed by prescribing physicians or qualified designees using the Martin Vigorimeter, measuring strength in kilopascals (kPa) ranging from 0 to 160 kPa.
Change From Screening in Bilateral Grip Strength | Screening, at 12, 24 and 54 weeks
  Bilateral hand grip strength assessments will be performed by prescribing physicians or qualified designees using the Martin Vigorimeter, measuring strength in kPa ranging from 0 to 160 kPa.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From start of study drug administration up to 54 weeks
Number of Participants With Infusion Discontinuations, Interruptions, and Infusion Rate Reductions due to TAK-411 Related TEAEs | From start of study drug administration up to 54 weeks
Number of Participants With Antibodies Against Host Cell Proteins (HCP), Beta-1,4-galactosyltransferase (B4GalT1) and Alpha-2,6-sialyltransferase (St6Gal1) | Up to 54 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (22):
- United States (15):
  - University of California San Diego, La Jolla, California
  - California Pacific Medical Center, San Francisco, California
  - UF Health Neurology - Jacksonville, Jacksonville, Florida
  - Visionary Investigators Network, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - The Curators of the University of Missouri on behalf of University of Missouri Health Care, Columbia, Missouri
  - The Washington University, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Penn Blood Disorders Program - Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Houston Methodist Research Institute, Houston, Texas
  - University of Washington, Seattle, Washington
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University Health Network, Toronto, Ontario
- Colombia (5):
  - Neuro ClinicaS.A.S, Medellín, Antioquia
  - Hospital Universitario San Ignacio, Bogotá, D.C.
  - Fundacion Valle del Lili, Cali, Valle del Cauca Department
  - Universidad del Rosario, Bogotá
  - Fundacion Oftalmologica de Santander - FOSCAL, Bucaramanga

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/95d6b5d68f4c4449??page=1&idFilter=TAK-411-2001